CLINICAL TRIAL: NCT03857308
Title: Eudaimonia and Sleep: Effects of a Mindfulness Intervention in Caregivers of People With Dementia
Acronym: CARING
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to continue enrollment for dissertation study due to COVID-19
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20011802
Record Dates: First submitted 2019-01-07; First posted 2019-02-27 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Caregivers; Burnout; Sleep
Keywords: well-being; sleep; caregiver
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training (Experimental)
  Interventions: Behavioral: Mindfulness Training
- Reappraisal Training (Active Comparator)
  Interventions: Behavioral: Reappraisal Training

INTERVENTIONS:
Behavioral: Mindfulness Training — This stress reduction training will last 14 days and teach participants skills in concentration, monitoring of present-moment bodily experience, and acceptance of experience. Participants are encouraged to "mentally welcome" all physical and emotional experience. Each day will consist of approximately 25 to 30 minutes of training.
  A full explanation of the mindfulness training compared to the reappraisal training could interfere with study blinding procedures. A complete description can be provided after data collection is complete.
  Arms: Mindfulness Training
Behavioral: Reappraisal Training — This stress reduction training will last 14-days. Each day consists of 25 to 30 minutes of daily practice in "Coping control." Participants are encouraged to reframe and reappraise life events, both past and present, and encouraged to solve personal problems through active change.
  A full explanation of the reappraisal stress reduction program compared to the mindfulness program could interfere with study blinding procedures. A complete description can be provided after data collection is complete.
  Other Names: My Time
  Arms: Reappraisal Training

SUMMARY:
This research study seeks to understand how stress reduction training influences caregiver well-being, sleep, and physiological responses to stress. All participants are caregivers of persons with dementia. Participants will complete a 14-day, online stress-reduction intervention which involves approximately 25-30 minutes of daily practice.

DETAILED DESCRIPTION:
The research project will be conducted over approximately 9 months and will consist of three data collection sessions for each participant. The three data sessions will occur before, after, and at 3-month follow-up of an 14-day, online stress-reduction training, in which participants will be asked to complete about 25 to 30 minutes of practice each day in one of two stress-reduction techniques. Participants will be randomly assigned to either a mindfulness training program or a reappraisal training program. The mindfulness training emphasizes mindfulness-based techniques to reduce stress and promote well-being, whereas the reappraisal training emphasizes cognitive strategies to change one's perception of the stressor as a way to reduce stress and promote well-being.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Self-reporting informal caregivers of persons with dementia

Exclusion Criteria:

* Self-reported major depressive disorder with psychotic features
* History of schizophrenia
* Bipolar disorder
* Uncorrected severe sensory impairments or chronic debilitating health problems that could hinder participating in the interventions
* Previous MBSR training or regular meditative practice within previous 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Change in Eudaimonic well-being | Baseline to 2-weeks (post-intervention), and 3-month follow-up
  54 item self-reported scale assessing change in eudaimonic well-being from pre to post-intervention. Will be assessed using the Scales of Psychologica Well-being (SPWB; Ryff & Keyes, 1995)
  1 = strongly disagree, 6 = strongly agree. This scale range applies for the 6 subscales, which can stand-alone, or be summed to obtain a total Eudaimonic Well-Being score. For this study, we are primarily interested in investigated changes over time of the summed score for eudaimonic well-being. Higher scores indicate higher eudaimonic well-being.
Change in Sleep Quality | Baseline to 2-weeks (post-intervention), and 3-month follow-up
  We will use a sleep diary that involves self-reported sleep habits, which we will use to calculate sleep onset, wake after sleep onset, and sleep efficiency. This will allow us to understand any changes in overall sleep quality across the intervention.
Change in Sleep Quality: Actigraph | Baseline to 2-weeks (post-intervention), and 3-month follow-up
  Actigraphic measure of limb movements used to calculate sleep efficiency, which is an assessment of the quality of sleep participants have.

SECONDARY OUTCOMES:
Change in Relationship Quality | Baseline to 2-weeks (post-intervention), and 3-month follow-up
  The Mutuality Scale of Family Care Inventory (Archbold, Stewart, Greenlick, & Harvath, 1990) will be used to assess for change in caregiver/care recipient relationship quality. It is a 15-item self-report measure to assess caregiver's perceived relationship quality with the care recipient. The scale items range in score from 1 to 4, with higher scores indicating greater relationship quality. Items are summed to create a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Dzierzewski, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States